CLINICAL TRIAL: NCT05620914
Title: A Window of Opportunity Study of Patritumab Deruxtecan in Patients With Brain Metastases
Acronym: PARAMETer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study sponsor, Daiichi, decided to close for mult reasons, including drug near expiration, lack of enrollment, and their priority changes.
Sponsor: Mustafa Khasraw, MBChB, MD, FRCP, FRACP (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor-Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Sponsor-Invesgitator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109490
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases, Adult
Keywords: Brain metastasis; Brain cancer; craniotomy; Patritumab Deruxtecan; Mustafa Khasraw; Pro00109490
MeSH Terms: conditions — Brain Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patritumab deruxtecan (Experimental): 15 participants with surgically-resectable brain metastases from multiple solid tumor primary histologies known to express HER3 will be treated. Patritumab deruxtecan (HER3-DXd) will be administered IV 5.6 mg/kg as a single dose 1-3 days prior to planned craniotomy and resection of BrM. Participants will undergo specimen collection prior to and during the planned craniotomy, including tumor, blood, and cerebrospinal fluid (CSF).
  Interventions: Drug: Patritumab deruxtecan

INTERVENTIONS:
Drug: Patritumab deruxtecan — Patritumab deruxtecan (HER3-DXd) will be administered IV 5.6 mg/kg as a single dose 1-3 days prior to planned craniotomy and resection of brain metastasis

SUMMARY:
The purpose of this study is to determine if the study drug, patritumab deruxtecan (HER3-DXd), can be measured in brain tumor tissue after recieving one dose of patritumab deruxtecan before surgery.

DETAILED DESCRIPTION:
This peri-operative window of opportunity study in patients with brain metastases will provide a single dose of the antibody-drug conjugate (ADC) patritumab deruxtecan (HER3-DXd, formerly U3-1402) prior to craniotomy to investigate pharmacokinetics, pharmacodynamics, intra- and peritumoral immune activation and responses, safety and explore potential biomarkers. This study will measure the level of the released payload DXd (MAAA-1181a) of patritumab deruxtecan, in resected brain metastasis (BrM) tissue.

Patients will receive a single dose of patritumab deruxtecan intravenously before surgery. Patients will also have procedures such as medical history review, blood draws, MRI scans, ECGs, and lumbar punctures. The amount of time patients are expected to be in this study is approximately 40 days.

Some of the risks of patritumab deruxtecan are diarrhea, nausea, vomiting, fatigue, headache, interstitial lung disease, and low blood counts.

All participants who are administered patritumab deruxtecan as part of this peri-operative window of opportunity study will be included in analyses summarizing adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have newly diagnosed or recurrent brain metastases, with one of the metastases being surgically resectable. Primary tumor histology must be one of the following solid tumor types:

   1. Melanoma (cutaneous skin)
   2. Stomach adenocarcinoma (intestinal subtype)
   3. Breast invasive carcinoma

      * ER+/PR+/HER2-
      * HER2+ (any ER/PR status)
      * Triple negative (ER-/PR-/HER2-)
   4. Colorectal adenocarcinoma
   5. Bladder Urothelial carcinoma
   6. Ovarian serous cystadenocarcinoma

      * Serous subtype
      * Mucinous subtype
   7. Cholangiocarcinoma
   8. Prostate adenocarcinoma
   9. Lung carcinoma

      * Non-small cell lung cancer (NSCLC)
      * Small cell lung cancer (SCLC)
2. Participant must be asymptomatic or minimally/well-controlled symptomatic from brain metastasis.

   1. Asymptomatic is defined as free of neurologic signs and symptoms related to metastatic brain lesions and not having required or received systemic corticosteroid therapy within 10 days prior to administration of patritumab deruxtecan.
   2. Minimally/well-controlled symptomatic is define as having neurologic signs and symptoms may be treated with a total daily dose of no more than 4 mg of dexamethasone (or equivalent) that is stable or tapering for 10 days prior to administration of patritumab deruxtecan. Participants with neurologic signs and symptoms who are not being treated with steroids are eligible and should have no experience of seizure within 10 days prior to administration of patritumab deruxtecan.
3. Participant must be willing and eligible for craniotomy.
4. Participant or partner(s) meets one of the following criteria:

   1. If the participant is a female of childbearing potential, she must have a negative serum pregnancy test at screening and must be willing to use a highly effective birth control, as detailed in Section 16.1.1, upon enrollment, during the Treatment Period, and for 7 months, following the last dose of study drug. A female is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy) with surgery at least 1 month before the first dose or confirmed by follicle stimulating hormone (FSH) test.
   2. Female participants must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.
   3. If male, the participant must be surgically sterile or willing to use a highly effective birth control (Section 16.1.1) upon enrollment, during the treatment period, and for at least 4 months following the last dose of study drug.
   4. Male participants must not freeze or donate sperm starting at screening and throughout the study period, and for at least 4 months after the final study drug administration.
5. Age ≥ 18 years of age at the time of entry into the study.
6. Karnofsky Performance Score (KPS) of 70 or higher.
7. Participants must have adequate bone marrow reserve and organ function, based on local laboratory data within 14 days prior to administration of patritumab deruxtecan, defined as:

   Laboratory Test Laboratory Value
   * Platelet count ≥100 000/mm3 or ≥100 × 109/L (platelet transfusions are not allowed up to 14 days prior to Cycle 1 Day 1 to meet eligibility)
   * Hemoglobin (Hgb) ≥9.0 g/dL (transfusion and/or colony stimulating factor support is allowed)
   * Absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5 × 109/L
   * Creatinine Clearance (CrCl) Creatinine clearance (CrCl) ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl;
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤3 × ULN (if liver metastases are present, ≤5 ×ULN)
   * Total bilirubin (TBL) ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases)
   * Serum albumin ≥2.5 g/dL
   * Prothrombin time (PT) or Prothrombin time- international normalized ratio (PT-INR) and activated partial thromboplastin time (aPTT)/partial thromboplastin time (PTT) ≤1.5 × (ULN), except for subjects receiving coumadin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator
8. A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Participants must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study
9. Ability to undergo MRI

Exclusion Criteria:

1. Female participants who are pregnant or breast-feeding or intend to become pregnant during the study.
2. Participants with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate.
3. Participants with severe, active co-morbidity, defined as follow:

   1. Participants with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C).
   2. Participants with known immunosuppressive disease or known human immunodeficiency virus (HIV) infection.
   3. Participants with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4).
4. Participants with another malignancy within 1 year prior, except for adequately resected non-melanoma skin cancer, superficial bladder tumors (Ta, Tis, T1), adequately treated intraepithelial carcinoma of the cervix uteri, low risk non-metastatic prostate cancer (With Gleason score <7 and following local treatment or ongoing active surveillance), curatively treated in-situ disease, or other solid tumors curatively treated.
5. Participants with a known history of hypersensitivity to patritumab deruxtecan, or any components of patritumab deruxtecan.
6. Participants who were previously treated with patritumab deruxtecan
7. Participants with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months.
8. Participants with any history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis), has current ILD, or is suspected to have such disease by imaging during screening.
9. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.)
10. Any autoimmune connective tissue or inflammatory disorders (e.g., Rheumatoid arthritis, Sjogren's, sarcoidosis, etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
11. Prior complete pneumonectomy
12. Participant is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
13. Evidence of any leptomeningeal disease.
14. Has clinically significant corneal disease.
15. Any evidence of severe or uncontrolled systemic diseases (including active bleeding diatheses, active infection, psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the Investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required for eligibility.
16. Inadequate washout period prior to Cycle 1 Day 1, defined as:

    1. Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days.
    2. Any cytotoxic chemotherapy, investigational agents or other anticancer drug(s) from a previous cancer treatment regimen or clinical study <14 days or 5 half-lives, whichever is longer.
    3. Monoclonal antibodies other than immune checkpoint inhibitors, such as bevacizumab (anti-VEGF) and cetuximab (anti-EGFR) <28 days.
    4. Immune checkpoint inhibitor therapy < 21 days.
    5. Major surgery (excluding placement of vascular access) < 28 days.
    6. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation < 28 days or palliative radiation therapy < 14 days.
    7. Chloroquine or hydroxychloroquine ≤ 14 days.
17. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, grade ≤1 or baseline. Participants with chronic, stable Grade 2 toxicities (defined as no worsening to > Grade 2 for at least 3 months prior to randomization/cycle 1 day 1 and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, comprised of:

    (a) Chemotherapy induced neuropathy (b) fatigue (c) residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include: (i) hypothyroidism/hyperthyroidism (ii) Type I diabetes (iii) hyperglycemia (iv) adrenal insufficiency (v) adrenalitis (vi) skin hypopigmentation (vitiligo)
18. Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day 1, including:

    1. QT interval corrected by Fridericia's formula (QTcF) prolongation interval of >450 ms (average of triplicate determinations at screening).
    2. Resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).
    3. Myocardial infarction within 6 months.
    4. New York Heart Association (NYHA) Classes 2 to 4 congestive heart failure within 28 days.
    5. Uncontrolled angina pectoris within 6 months.
    6. Cardiac arrhythmia requiring antiarrhythmic treatment.
    7. Left ventricular ejection fraction (LVEF) <50%
19. Active Hepatitis B and/or Hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1, Day 1.

    a) Participants with past or resolved Hepatitis B virus (HBV) infection are eligible if: i) Hepatitis surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) positive; OR ii) HBsAg positive and HBV DNA viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases (in the absence of liver metastasis); OR iii) HBsAg positive and HBV DNA viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with liver metastasis and abnormal transaminases AST/ALT < 3 ULN.

    b) Participants with a history of Hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection, is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (ie, sustained viral response according to the local product label but no less than 12 weeks, whichever is longer).
20. Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's judgment, could affect the safety of the subject; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results
21. Subjects with human immunodeficiency virus (HIV) infection.
22. Has known hypersensitivity to either the drug substance or inactive ingredients in the drug product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Determine the concentration of DXd in brain metastasis tumor tissue after one dose of the HER3-targeted ADC patritumab deruxtecan (HER3-DXd) administered via IV 1-3 days prior to craniotomy. | 3 days
  The mean concentration of the DXd payload from patritumab deruxtecan will be computed. In addition, the distribution of the concentration will be examined

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of ADC in serum, including ADC concentration and DXd concentration, collected at screening, pre-infusion, post-infusion, 4 hours post-infusion, 24 hours after patritumab deruxtecan administration, and at craniotomy. | 3 days
  Changes between screening and each follow-up assessment in pharmacokinetics measures will be computed. All patients who have at least one post-infusion serum sample will be included in these analyses.
Assess the evidence of tumor cell death via histopathological examination and measurement of γH2AX levels in tumor tissue. | 3 days
  Among those patients who have an evaluable Brain Met tissue, the level of γH2AX in the resected BrM tissue will be described with means, standard deviations, and other statistics if needed.
Assess the safety of patritumab deruxtecan in patients with brain metastasis after the single dose and up to 40+7 days. | 40 days
  The proportion of patients who experience each type of adverse event will be tabulated by the maximum grade experienced. The first summary will reflect all adverse events; whereas the second summary will reflect only adverse events that are possibly, probably, or definitely related to treatment with patritumab dereuxtecan.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials